CLINICAL TRIAL: NCT02271906
Title: The ATTAIN Study: A Therapeutic Trial of Afatinib In the Neoadjuvant Setting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0305; NCI-2015-00357 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non small cell lung cancer; NSCLC; Adenocarcinoma; Squamous cell carcinoma; BIBW 2992; Afatinib
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIBW 2992 (Experimental): BIBW 2992 40 mg by mouth daily for a minimum of 14 days, and until the day of surgery.
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — 40 mg by mouth daily for a minimum of 14 days, and until the day of surgery.

SUMMARY:
The goal of this clinical research study is to learn if it is tolerable for patients with NSCLC to receive afatinib before surgery. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take afatinib by mouth 1 time a day for at least 14 days before your surgery. You should take it at least 1 hour before or 2 hours after a meal. You will sign a separate consent form that describes the surgery and its risks in more detail.

You will keep a diary of when you take the pills. You should bring the diary to each visit, along with your pill bottle so the study staff can count any remaining pills.

Some side effects, such as diarrhea and skin rash, will occur in almost all patients. If you have severe side effects, your dose may be lowered.

Study Visits:

One (1) time a week while you are taking afatinib:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.

Within a week before your surgery:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a PET-CT scan to check the status of the disease.
* You will have a MUGA scan to check your heart function.

On the day of surgery, blood (about 3 teaspoons) will be drawn for research tests, including looking for tumor cells that may be in the blood.

Leftover tissue from surgery will be used for biomarker testing.

Length of Treatment:

You will take your last dose of study drug within 24 hours before your surgery. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visit.

Follow-Up:

At about 30 days after surgery:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.

It is possible that the study staff will call you instead of the visit above. You will be asked how you are doing. The call should last about 5 minutes.

If you are having side effects from the study drug at the time of the follow-up visit or call, you may have additional follow-up if the doctor thinks it is needed. The follow-up tests, procedures, and schedule will be the doctor's decision depending on the side effects.

This is an investigational study. Afatinib is FDA approved and commercially available to be the first treatment for patients with a specific type of NSCLC that has spread. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC, who are deemed to be surgical candidates by standard criteria. Patients with all types of NSCLC (e.g., adenocarcinoma, squamous cell carcinoma) will be allowed to enroll.
2. Patients with Stage IA to IIB disease. Select patients with resectable stage IIIA disease (T3N1, T4N0, T4N1) will also be eligible if approved by the PI.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
4. Measurable disease by RECIST 1.1 criteria
5. Mediastinoscopy and/or Endoscopic Bronchial Ultrasound (EBUS) and/or Endoscopic Ultrasound (EUS) for complete surgical staging when clinically indicated
6. Serious, active infections must be controlled. Patients may be enrolled while still on antibiotics as long as clinical signs of active infection have resolved.
7. A signed informed consent document (ICD)
8. Patients 18 years or older
9. Able and willing to take oral medications

Exclusion Criteria:

1. Known preexisting interstitial lung disease, interstitial pulmonary fibrosis, or connective tissue disorder associated lung disease
2. Known N2 nodal disease or distant metastatic disease
3. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomization.
4. Patients with any of the following lab values at screening should be excluded: Absolute neutrophil count (ANC) < 1500 / mm^3; Platelet count < 100,000 / mm^3; Serum creatinine >/= 1.5 times the upper normal limit or calculated/measured creatinine clearance </= 60 mL/min; Bilirubin >/=1.5mg/dL (> 26 mol/L, SI unit equivalent); Aspartate amino transferase (AST) or Alanine amino transferase (ALT) >/= three (3) times the upper limit of normal.
5. Active hepatitis B infection, active hepatitis C infection or known HIV carrier.
6. Known or suspected active drug or alcohol abuse
7. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom for example Crohn's disease, malabsorption or CTC grade >/= 2 diarrhea of any etiology.
8. Baseline (< 1 month before treatment) cardiac left ventricular function with resting ejection fraction of less than 50% measured by multigated blood pool imaging of the heart (MUGA scan) or echocardiogram
9. Patients receiving other investigational agent.
10. History of allergic reactions to anilinoquinazolins like gefitinib, erlotinib, or BIBW2992
11. Uncontrolled intercurrent illness that would preclude a patient from undergoing surgery
12. Psychiatric illness/social situations that would limit compliance with study requirements
13. Pregnant (positive pregnancy test) or lactating
14. Inability to comply with study and/or follow-up procedures
15. Patients who are not surgical candidates or refuse surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Simon, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two patients with untreated resectable Stage IA to IIIA non-small cell lung cancer were recruited at the University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Following registration, patients should begin protocol treatment within 2 weeks. If a patient does not receive protocol therapy within 2 weeks following registration, the patient's registration on the study may be canceled at the discretion of the study investigators and the patient will be considered a screen failure.
Groups:
- Afatinib Single Agent: Afatinib 40mg orally daily until day of surgery for a minimum of two weeks
Period: Overall Study
Arm/Group | Afatinib Single Agent
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib Single Agent
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 62 [49 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment "Completed"
Description: A patient is declared to have the treatment "completed" if he completes at least 14 days of neoadjuvant treatment, had a thoracotomy for the planned surgical resection, and 30 days of post operative care.
Time Frame: From the start of neoadjuvant treatment to 30 days post operative care
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib Single Agent
Number analyzed (Participants) | 2
Participants
  Treatment Completed | 2
  Treatment Not Completed | 0

2. Secondary Outcome: Number of Participants With a Change in Standard Uptake Value (SUV) From Pre to Post Operative PET-CT
Description: To determine whether pre-operative Afatinib treatment affects metabolic tumor labeling, as measured by PET-CT scanning.
Time Frame: From the start of neoadjuvant treatment to follow-up, up to 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib Single Agent
Number analyzed (Participants) | 2
Participants
  Increase in percentage change | 1
  Decrease in percentage change | 1

ADVERSE EVENTS:
Time Frame: From the start of neoadjuvant treatment to 30 days post operative care
Description: The grades 1-3 adverse events which were recorded after registration were included
Arm/Group | Afatinib Single Agent
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afatinib Single Agent (N=2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT02271906/Prot_SAP_000.pdf